CLINICAL TRIAL: NCT02687022
Title: A Comparative Study of Measurement Repeatability for Two Aberrometers
Brief Title: Measurement Repeatability in Contemporary Aberrometry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Bruce Allan, Consultant Ophthalmic Surgeon, Moorfields Eye Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ALLB1019
Record Dates: First submitted 2016-02-07; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Myopia (Peramis) (Experimental): Peramis aberrometry: 30 consecutive LASIK candidates with myopia and regular astigmatism who agree to participate in the study will have up to 4 aberrometry scans acquired consecutively using the Peramis (test) aberrometer.
  Interventions: Device: Peramis aberrometry
- Myopia (iDesign) (Active Comparator): iDesign aberrometry: The same 30 consecutive LASIK candidates scanned in the Myopia (Peramis) arm will also have up to 4 aberrometry scans acquired consecutively using the iDesign aberrometer (control) aberrometer. The order of scans (Peramis and iDesign) will be randomised.
  Interventions: Device: iDesign aberrometry
- Irregular astigmatism (Peramis) (Experimental): Peramis aberrometry: 30 consecutive cases with stage II-III keratoconus or post corneal transplantation cases with irregular astigmatism will have up to 4 aberrometry scans acquired consecutively using the Peramis (test) aberrometer
  Interventions: Device: Peramis aberrometry
- Irregular astigmatism (iDesign) (Active Comparator): iDesign aberrometry: 30 consecutive cases with stage II-III keratoconus or post corneal transplantation cases with irregular astigmatism will also have up to 4 aberrometry scans acquired consecutively using the iDesign aberrometer (control) aberrometer. The order of scans (Peramis and iDesign) will be randomised.
  Interventions: Device: iDesign aberrometry

INTERVENTIONS:
Device: Peramis aberrometry — A non-invasive photographic scan sequence acquired in under 10 seconds
  Other Names: Wavefront scanning
  Arms: Irregular astigmatism (Peramis); Myopia (Peramis)
Device: iDesign aberrometry — A non-invasive photographic scan sequence acquired in under 10 seconds
  Other Names: Wavefront scanning
  Arms: Irregular astigmatism (iDesign); Myopia (iDesign)

SUMMARY:
Wavefront scans are a common form of diagnostic test applied in preparing patients for laser eye surgery. An optical map of the eye is created by wavefront scanning, and information from these maps is used to program lasers used to correct focusing errors in the eye. Here the investigators are comparing how repeatable measurements are with a new wavefront scanner and one that is already in widespread use.

DETAILED DESCRIPTION:
Aberrometers are used to measure each element of defocus (aberration) in an optical system. In LASIK, information derived from aberrometry (scans performed using aberrometers) is used to program the pattern of laser pulses delivered by an excimer laser in therapeutic reshaping of the cornea to correct defocus. To do this accurately, aberrometry findings need to be repeatable and correspond closely to manifest refraction. Here the investigators compare repeatability of measurements for a new aberrometer (Peramis) versus the aberrometer most widely used in contemporary wavefront guided laser vision correction (iDesign).

The test aberrometer will be:

Peramis (Schwind Eye-tech Solutions, Kleinostheim, Germany).

Control aberrometer will be:

iDesign (AMO, Santa Clara, CA)

ELIGIBILITY:
Inclusion Criteria:

* Myopic LASIK candidates (manifest refraction spherical equivalent range 0 to -10 diopters with up to 6 diopters cylinder) or patients attending corneal service with stage II-III keratoconus or post-keratoplasty

Exclusion Criteria:

* Visually significant co-pathology (CDVA<6/6) other than irregular astigmatism;
* Patients unable to complete a sequence of 2 good scans (acquisition diameter >5mm) in one eye within 4 attempts

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
2nd to 4th order aberrations (5mm pupil). | <10 seconds
  M, J0, J45, Coma, Trefoil, Spherical Aberration. Different types of defocus or aberration can be defined and measured by wavefront scanning. Aberrations are classified and quantified by a mathematical treatment called Zernike analysis in which harmonic elements of the waveform of the light detected by the wavefront sensor (aberrometer) are quantified in sequence, starting with simple (lower order) waveforms such as sphere and cylinder (M, J0, J45) corrected in a normal spectacle prescription, and progressing through more complex (higher order) waveforms including, coma, trefoil and spherical aberration which may influence quality of vision. The amount of each aberration varies as a function of pupil size. So pupil size is standardised at 5mm diameter for quantification.

SECONDARY OUTCOMES:
% of patients with qualifying scan sequence | <5 minutes
  % of patients in whom two 5mm diameter aberrometry scans can be acquired within 4 attempts

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Allan, MD FRCOphth, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to publish summary descriptive data and analyses. Anonymised individual data will be available to systematic reviewers on request.

REFERENCES:
- [Background] Visser N, Berendschot TT, Verbakel F, Tan AN, de Brabander J, Nuijts RM. Evaluation of the comparability and repeatability of four wavefront aberrometers. Invest Ophthalmol Vis Sci. 2011 Mar 10;52(3):1302-11. doi: 10.1167/iovs.10-5841. PMID 21051697
- [Background] LeDue J, Jolissaint L, Veran JP, Bradley C. Calibration and testing with real turbulence of a pyramid sensor employing static modulation. Opt Express. 2009 Apr 27;17(9):7186-95. doi: 10.1364/oe.17.007186. PMID 19399094
- [Background] Cagigal MP, Valle PJ. Wavefront sensing using diffractive elements. Opt Lett. 2012 Sep 15;37(18):3813-5. doi: 10.1364/ol.37.003813. PMID 23041868
- [Background] Jung JW, Chung BH, Han SH, Kim EK, Seo KY, Kim TI. Comparison of Measurements and Clinical Outcomes After Wavefront-Guided LASEK Between iDesign and WaveScan. J Refract Surg. 2015 Jun;31(6):398-405. doi: 10.3928/1081597X-20150521-06. PMID 26046707